CLINICAL TRIAL: NCT05380362
Title: Prospective Randomized Endovascular Therapy in Multiple Sclerosis
Acronym: PREMiSe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Volcano Corporation (Industry)
Responsible Party: Principal Investigator, Adnan H. Siddiqui, MD, PhD, Associate Professor of Neurosurgery and Radiology, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PREM 01; NSG1730210B (Other: HSIRB - SUNY Buffalo)
Record Dates: First submitted 2013-04-17; First posted 2022-05-18 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Venous Angioplasty (Experimental): 20 patients will have venous angio plasty
  Interventions: Other: Venous Angioplasty
- Angio with no plasty (Sham Comparator): Patients will be brought to the angio suite and given and angio but no plasty although patient will not be aware of which treatment they are having.
  Interventions: Other: Sham Angioplasty

INTERVENTIONS:
Other: Venous Angioplasty — venous angiogram to look for lesions or flaps and then plastying vessels open.
  Arms: Venous Angioplasty
Other: Sham Angioplasty — Patients will be brought to the angio suite and will not know if they are having the venous angioplasty or not.
  Arms: Angio with no plasty

SUMMARY:
1. To assess the safety of endovascular therapy (balloon angioplasty) for venous stenoses in MS patients with CCSVI as documented by sonographic (extracranial echocolor-Doppler (ECD) and transcranial color Doppler (TCD)
2. To study the morphology of the venous anomalies by using intraluminal ultrasound (IVUS).
3. To evaluate preliminary efficacy of endovascular therapy (angioplasty) as measured by clinical (relapse rate, disability progression (EDSS)), sonographic (ECD/TCD) and MRI/MRV parameters.
4. To evaluate change in patients self-reported QOL following the therapeutic angioplasty
5. To evaluate whether changes in QOL, fatigue, MSFC or attention following therapeutic angioplasty are associated with brain changes as measured by functional MRI (fMRI).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years

  * EDSS 0-6.5
  * Diagnosis of relapsing MS according to the McDonald criteria (Polman et al., 2005)
  * Be on treatment with currently FDA approved disease-modifying treatments
  * Evidence of ≥2 sonographic parameters of suspicious abnormal extracranial cerebral venous outflow (see Table 1 background and 1.5 section)
  * Demonstration of venous occlusive disease on cervical MRV
  * Normal renal function: creatinine clearance level of >60:

Constant= 1.23 for men; 1.04 for women

Exclusion Criteria:

* • Relapse, disease progression and steroid treatment in the 30 days preceding study entry

  * Pre-existing medical conditions known to be associated with brain pathology (e.g., neurodegenerative disorder, cerebrovascular disease, positive history of alcohol abuse, etc.)
  * Severe peripheral chronic venous insufficiency
  * Abnormal renal function
  * Contrast allergy (anaphylaxis)
  * Not accepting to undergo the endovascular treatment
  * Peripheral Vascular Disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adnan H Siddiqui, M.D., Ph. D., Principal Investigator — University at Buffalo Neurosurgery
Locations (1):
- Gates Circle Hospital, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Venous Angioplasty | Angio With no Plasty
Started | 10 | 10
Completed | 9 | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Venous Angioplasty | Angio With no Plasty | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (8.2) | 44.8 (10.5) | 44.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 4 | 2 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Immediate and Short-term SAE
Description: Percent (%) of patients with Severe Adverse Events (SAE) measured at 1 month (Short term) post-surgical safety outcome in MS patients diagnosed with CCSVI that underwent therapeutic angioplasty. The 95% confidence interval of the SAE rates for immediate and short terms will be obtained by the exact method, respectively. The immediate and short term SAE rates will be analyzed, respectively, using the Fisher's exact test.
Time Frame: 1 month post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Venous Angioplasty | Angio With no Plasty
Number analyzed (Participants) | 9 | 10
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Venous Angioplasty | Angio With no Plasty
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 3/9 | 3/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Venous Angioplasty (N=9) | Angio With no Plasty (N=10)
Immune thrombocytopenic purpura (Immune system disorders) | 0 | 1 — Immune thrombocytopenic purpura treated with 100mg prednisone once daily
Bladder infection (Renal and urinary disorders) | 0 | 1 — Bladder infection treated with antibiotics over 10 days
Shingles (Nervous system disorders) | 0 | 1 — Diagnosis of shingles treated with Valtrex (GlaxoSmithKline) 3x daily for 7 days
Cardiac event (Cardiac disorders) | 1 | 0 — Cardiac event treated with pacemaker installation
Swelling & Soreness (General disorders) | 1 | 0 — Swelling and soreness at left side of the neck, no treatment required
Transobturator sling (Renal and urinary disorders) | 1 | 0 — Hospitalization for scheduled transobturator sling procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No